CLINICAL TRIAL: NCT05043532
Title: Randomized Trial to Evaluate the Optimal Number of Passes Required for Molecular Profiling During Endoscopic Ultrasound-guided Fine Needle Biopsy of Pancreatic Adenocarcinoma
Brief Title: Randomized Trial for Optimal Number of Passes Required for Molecular Profiling During EUS-FNB of Pancreatic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 21.069.05; 1741103 (Other: Orlando Health IRB)
Record Dates: First submitted 2021-09-07; First posted 2021-09-14 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer; Pancreatic Neoplasms; Adenocarcinoma of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient undergoing the procedure, research coordinator calling patients for follow-up and the pathologist performing molecular profiling will be blinded to the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two passes performed during EUS-FNB of pancreatic adenocarcinoma (Active Comparator): Once the pancreatic mass is identified on endoscopic ultrasound examination, total of two passes will be performed during find needle biopsy and placed in 10% formalin for processing for molecular profiling.
  Interventions: Procedure: 2 passes during EUS-guided fine needle biopsy
- Three passes performed during EUS-FNB of pancreatic adenocarcinoma (Active Comparator): Once the pancreatic mass is identified on endoscopic ultrasound examination, total of three passes will be performed during find needle biopsy and placed in 10% formalin for processing for molecular profiling.
  Interventions: Procedure: 3 passes during EUS-guided fine needle biopsy

INTERVENTIONS:
Procedure: 2 passes during EUS-guided fine needle biopsy — Once the pancreatic mass has been visualized on endoscopic ultrasound, a total of two passes will be performed and placed in 10% formalin for processing for molecular profiling. Onsite evaluation will be performed using a part of the sample from the first pass in order to establish onsite diagnostic adequacy in all patients.
  Arms: Two passes performed during EUS-FNB of pancreatic adenocarcinoma
Procedure: 3 passes during EUS-guided fine needle biopsy — Once the pancreatic mass has been visualized on endoscopic ultrasound, a total of three passes will be performed and placed in 10% formalin for processing for molecular profiling. Onsite evaluation will be performed using a part of the sample from the first pass in order to establish onsite diagnostic adequacy in all patients.
  Arms: Three passes performed during EUS-FNB of pancreatic adenocarcinoma

SUMMARY:
This is a randomized trial to evaluate the optimal number of passes required during endoscopic ultrasound-guided fine needle biopsy for molecular profiling in pancreatic cancer

DETAILED DESCRIPTION:
Endoscopic ultrasound-guided fine needle tissue acquisition is currently the gold standard for sampling solid pancreatic masses. By using novel fine needle biopsy (FNB) needles during EUS-guided tissue sampling, core tissue samples can also now be obtained, with diagnostic adequacy of >90%.

Molecular profiling is becoming increasingly important in the management of pancreatic adenocarcinoma for targeted therapy. As the procurement of core tissue is possible with EUS-FNB, adequate tissue can now be obtained for molecular profiling. However, the number of passes required during EUS-FNB to obtain sufficient quantity of core tissue to successfully perform molecular profiling is unknown, although usually 2-3 passes are performed as standard of care practice.

The primary aim of this study is therefore to elucidate the optimal number of passes required during EUS-FNB to procure adequate tissue for molecular profiling in patients with pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and over
2. Suspected or confirmed pancreatic mass seen on imaging, requiring endoscopic ultrasound-guided fine needle biopsy

Exclusion Criteria:

1. Age < 18 years
2. Females who are pregnant
3. Pancreatic mass is not accessible for fine needle biopsy via endoscopic ultrasound
4. Biopsied pancreatic mass is not adenocarcinoma on pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of ability to perform successful molecular profiling in core tissue obtained during EUS-guided fine needle biopsy | 7 days
  Rate of ability to perform successful molecular profiling in core tissue obtained during EUS-guided fine needle biopsy of pancreatic adenocarcinoma, with comparison between two and three passes during fine needle biopsy

SECONDARY OUTCOMES:
Number of actionable mutations detected on molecular profiling | 7 days
  Number of actionable mutations detected on molecular profiling
Rate of technical success | 1 day
  Rate of technical success of EUS-guided fine needle biopsy. Technical success is defined as the successful completion of the EUS-guided fine needle biopsy procedure.
Rate of procedure-related adverse events | 7 days
  Rate of procedure-related adverse events, defined as any adverse event occurring as a result of EUS-guided fine needle biopsy
Type of actionable mutations detected on molecular profiling | 7 days
  Type of actionable mutations detected on molecular profiling

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Bang, MD MPH, Principal Investigator — Orlando Health
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No